CLINICAL TRIAL: NCT01445483
Title: A Pilot Study to Evaluate Neuropsychological Outcome Measures and Their Relationship With Prognosis in Patients Receiving Radiation Therapy for Brain Metastases
Brief Title: Neuropsychological Changes in Patients Receiving Radiation Therapy for Brain Metastases
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080214; 08-C-0214; NCT00769444 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-06-26

CONDITIONS: Brain Metastasis; Cancer
Keywords: Cancer; Radiation; Brain; Neuropsychological Outcome; Metastasis; Natural History; Brain Metastasis
MeSH Terms: conditions — Brain Neoplasms; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1/Cohort 1: KPS>70; Age =65; controlled primary tumor and no extracranial metastases
- 2/Cohort 2: KPS>70 and at least one of the following: age >65, uncontrolled or synchronous primary disease, or extracranial metastases
- 3/Cohort 3: KPS<70

SUMMARY:
Background:

* There are no standardized sets of tests to measure changes in neuropsychological functioning in patients treated for brain metastasis (cancer that has spread beyond the original site to the brain).
* Neuropsychological function has an important effect on quality of life and should be included when determining treatment options.

Objectives:

* To find out if there is a change in patients cognitive (thinking) and daily functioning after standard radiation treatment for brain metastasis that can be measured with tests.
* To see if any changes on these tests are related to patients response to radiation therapy.

Eligibility:

- Patients 18 years of age or older who have cancer that has spread to the brain.

Design:

* Patients receive a 2-week course of radiation therapy to the brain, given daily 5 days a week. Some patients may require stereotactic radiosurgery (an additional boost of radiation therapy to specific sites of brain metastasis).
* Patients have the following evaluations before and after treatment to determine changes in cognition and functioning:
* Neuropsychological testing to measure cognitive (thinking) abilities like memory, attention, processing speed, and reading, and fine motor skills.
* Questionnaires to assess quality of life and daily living skills.
* Patients have MRI scans and blood and urine tests.
* At the completion of radiation treatment, patients return to the clinic for follow-up visits at 1, 2, 4, 6, 9 and 12 months for blood and urine tests, physical examination, MRI of the brain, neuropsychological testing and assessments of quality of life and daily living skills.

DETAILED DESCRIPTION:
Background:

* Metastatic brain tumors occur more frequently than primary brain tumors and occur in approximately 25 percent of patients who die of cancer each year.
* The Radiation Therapy Oncology Group (RTOG) developed three prognostic classes using a recursive partitioning analysis (RPA) of a large database. These classes are based on Karnofsky Performance Status (KPS), age and disease status.
* The RTOG RPA classes do not include neuropsychological function as a measure of outcome.
* There is no consensus of standardization of test selection to measure changes in neuropsychological functioning in this patient population.
* Neuropsychological function has an important effect on quality of life and should be included when determining prognosis and treatment options for patients.
* Neuropsychological functioning is important when determining the effects of treatments and for measuring outcomes in clinical trials.

Objectives:

* To identify the neuropsychological test scores which detect significant change in neuropsychological functioning in patients receiving radiation therapy for brain metastases.
* To examine the relationship between neuropsychological function and survival in patients receiving radiation therapy for brain metastases.

Eligibility:

* Patients aged 18 years and older.
* Pathologically confirmed primary malignancy with at least one intraparenchymal brain metastasis as identified on brain MRI scan with intravenous contrast.
* The patient must communicate in English in order to complete the neuropsychological evaluations.

Design:

* This is a longitudinal study that will administer serial neuropsychological assessments to patients with brain metastases who receive radiation therapy.
* Patients will undergo a battery of neuropsychological tests prior to radiotherapy (WBRT or WBRT followed by SRS), 2 weeks after completion of radiation therapy, then every 3 months for up to 12 months.
* The test battery will involve approximately 40 minutes of direct cognitive testing and 15 minutes of questionnaires.

There will be three cohorts of 20 patients each for a total of 60 patients. The three cohorts will be made up of differing histologies and will be sorted on the basis of their RTOG RPA Class.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients must be 18 years of age or older.
2. Pathologically confirmed primary malignancy with at least one intraparenchymal brain metastasis as identified on brain MRI scan with intravenous contrast.

   * Cohort 1 (N=20): KPS greater than 70; Age less than or equal to 65; controlled primary tumor and no extracranial metastases.
   * Cohort 2 (N=20): KPS greater than 70 and at least one of the following: age greater than 65, uncontrolled or synchronous primary disease, or extracranial metastases
   * Cohort 3 (N=20): KPS less than 70
3. Patient must have a primary medical or surgical oncologist in the community or at NCI who is willing to collaborate with the ROB staff in the clinical management of the patient.
4. All patients must sign a document of informed consent indicating their understanding of the investigational nature and the risks of this study BEFORE any of the protocol related studies are preformed (this does not include routine laboratory tests or imaging studies required to establish eligibility).
5. Subjects of childbearing or child- fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.

EXCLUSION CRITERIA:

1. Cognitively impaired patients who cannot give informed consent, including patients assigned a power of attorney for medical decisions.
2. Inability to communicate in the English language.
3. Pre- existing or active psychiatric or neurologic impairments, not caused by the brain metastasis, which, in the opinion of the investigators, will interfere with the proper administration or completion of the protocol.
4. Prior Therapy

   * Patients must not have been treated for a previous brain metastasis.
   * Patients must not have had previous cranial radiation.
   * Patients must not undergo treatment with an investigational drug for the primary disease within 7 days of baseline neuropsychological testing.
   * Patients must not receive systemic therapy within 7 days prior to baseline neuropsychological testing.
   * Patients who have had surgery for their current brain metastasis must wait at least 7 days before baseline neuropsychological testing.
5. Concurrent Therapy

   * Treatment of primary malignancy with systemic therapy (chemotherapy or biologic agents) cannot be delivered concurrently with the treatment of the intracranial disease. However, treatment of the primary site with local therapy, either surgery or radiotherapy, can be performed concurrently with the treatment of the intracranial disease.
   * Patients receiving glucocorticoids should be tapered to the lowest possible dose, or stopped altogether, by the treating physician. If glucocorticoid dose is adjusted or given for the first time, the patient must remain on stable dose of glucocorticoids for at least 24 hours prior to initial neurocognitive testing, CT and MR imaging.
6. Patients needing emergent radiation therapy for their brain metastases will be excluded.
7. Patients must not have evidence of leptomeningeal metastases.
8. Patients must not be HIV positive.
9. Other medical conditions deemed by the PI or associates to make the patient ineligible for protocol investigations.
10. Pregnant or breast-feeding females are excluded because of the potential mutagenic effects on a developing fetus or newborn.
11. Clinically significant unrelated systemic illness which in the judgment of the Principal or Associate Investigator would compromise the patient s ability to tolerate this therapy or are likely to interfere with the study procedures or results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-04-17 (Actual)

PRIMARY OUTCOMES:
Neuropsychological function | Completion of study
  To examine the relationship between neuropsychological function and survival in patients receiving radiation therapy for brain metastases
Test scores for: Hopkins Vrbl Learning Test recall; WAIS-III Digit Span; the WAIS-III Symbol Search; the Ruff 2 & 7 Selective Attn. The Trailmaking Tst Part B speed z-score; and the Grooved Pegboard Test dominant hand z-score | Completion of study
  To identify the neuropsychological test scores which detect significant change in neuropsychological functioning in patients receiving radiation therapy for brain metastases

SECONDARY OUTCOMES:
Strengths and weaknesses in neuropsychological functioning | completion of study
  To examine the strengths and weaknesses in neuropsychological functioning of patients with brain metastases after radiation therapy
RTOG RPA classification | completion of study
  To examine the relationship between the RTOG RPA classification for brain metastasis survival and baseline neuropsychological functioning
North American Adult Reading Test-Short Form (NART-35), Hopkins Verbal Learning Test (HVLT), WAIS-III Digit Span subtest, WAIS-III Symbol Search subtest, Ruff 2 and 7 Selective Attention Test | completion of study
  To further examine whether other measures from the following battery detect significant change in neuropsychological function or predict prognosis in this patient population
Neuropsychological functioning, brain lesions (e.g., number and volume), MRI abnormalities, biomarkers, and disease progression or recurrence | completion of study
  To investigate the relationship between neuropsychological functioning, brain lesions (e.g., number and volume), MRI abnormalities, biomarkers, and disease progression or recurrence
Neuropsychological functioning | completion of study
  To explore the neuropsychological functioning of patients with brain metastases treated with different therapies (e.g. chemotherapy, corticosteroids, complete surgical resection)
neuron specific enolase (NSE), S100B, MMPs and VEGF | completion of study
  To investigate the role of biomarkers, including neuron specific enolase (NSE), S100B, MMPs and VEGF as potential markers of brain injury and disease progression in the serum, plasma and urine of patients with brain metastases
Baseline neuropsychological data | completion of study
  To gather baseline neuropsychological data on patients with brain metastases for use as a reference in the development of new clinical trials involving this patient population in the ROB

CONTACTS AND LOCATIONS:
Overall Officials: DeeDee K Smart, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Johnson JD, Young B. Demographics of brain metastasis. Neurosurg Clin N Am. 1996 Jul;7(3):337-44. PMID 8823767
- [Background] Posner JB. Management of brain metastases. Rev Neurol (Paris). 1992;148(6-7):477-87. PMID 1448668
- [Background] Wen PY, Loeffler JS. Brain metastases. Curr Treat Options Oncol. 2000 Dec;1(5):447-58. doi: 10.1007/s11864-000-0072-3. PMID 12057152
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0214.html